CLINICAL TRIAL: NCT03906838
Title: Does Regional Anesthesia Reduce Postoperative Opioid Consumption in Subjects Undergoing Fibula Free Flap Reconstruction of the Head and Neck: A Prospective Trial
Brief Title: Regional Anesthesia Block in Fibula Free Flap Reconstruction
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: funding not obtained
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201900883
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Local; Surgery; Opioid Use; Pain, Postoperative; Head and Neck Neoplasms
MeSH Terms: conditions — Pain, Postoperative; Head and Neck Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regional Nerve Block (Experimental): Subjects in the regional anesthesia cohort will have a regional anesthesia block and/or catheter placement administered according to current hospital policies and our established standard of care.
  Interventions: Drug: Ropivacaine injection
- No Regional Nerve Block (No Intervention): Subjects in the no regional anesthesia cohort will not get pre-operative regional anesthesia, and their surgery and anesthesia will be performed according to normal policies and standard of care in our hospital.

INTERVENTIONS:
Drug: Ropivacaine injection — Regional Anesthesia Nerve Block: Incremental injections up to total of 20 mL of 0.5% ropivacaine is administered.
  Arms: Regional Nerve Block

SUMMARY:
Despite many recent advances in pain management, post-operative pain is widely considered to be poorly managed. Furthermore, the mainstay of current pain management is opioids, for which there is strong evidence of ill effects and long-term potential for addiction. There are many studies demonstrating that perineural regional anesthesia can be superior to intravenous opioid analgesia, and that the technique is safe. By using temporary implanted catheters, this method can now deliver prolonged analgesia, thus reducing the need for opioids in the postoperative period. Regional anesthesia is a proven technique and used daily by anesthesiologists, and it is also the first choice for hip and knee replacement surgery for orthopedic surgeons. Patients undergoing head and neck reconstruction with the use of free tissue transfer experience a significant amount of post-operative pain due to the complexity of the surgery, the presence of a head and neck surgical site as well as a secondary donor site, and existing co-morbidities, most commonly malignancy, that also cause significant pain. These patients often require opioids for pain control throughout the hospital stay, and are almost always discharged home with additional opioids. By utilizing regional anesthesia blocks at the donor sites, the investigators can potentially reduce post-operative pain while also reducing the use of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing microvascular fibula free flap reconstruction of the head and neck
* Subjects undergoing primary or secondary reconstruction

Exclusion Criteria:

* Subjects needing elevation of care to the intensive care unit due to remaining intubated for extended period of time or other complications during the peri or post operative period
* Subjects with surgical complications requiring significant alteration of the treatment plan

  o Subjects requiring a return to the operating room during admission will be excluded, unless it is for a procedure not related to the original surgery occurring after post op day 3, such as a gastrostomy tube or long term IV access.
* Subjects with true allergies to the study drugs
* Subjects undergoing reconstruction with more than 1 free flap, or with the use of any additional regional flaps
* History of substance dependence or enrollment in a pain management program
* Any subject currently enrolled in pain management, or currently taking long acting opioids such as methadone or oxycontin.
* Subjects who do not stay in the hospital for at least 4 days post operatively
* Subjects requiring anticoagulation will not require modifications prior to receiving regional anesthesia.
* Inability to properly place catheter or administer the regional anesthesia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 72 hours (3 days) post-operatively
  Defined by the research team as the subjects' morphine equivalent dose at 72 hours (3 days) post-operatively. The postoperative period commences at extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Fernandes, MD, DMD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Background] Werner MU, Soholm L, Rotboll-Nielsen P, Kehlet H. Does an acute pain service improve postoperative outcome? Anesth Analg. 2002 Nov;95(5):1361-72, table of contents. doi: 10.1097/00000539-200211000-00049. No abstract available. PMID 12401627
- [Background] Gwira Baumblatt JA, Wiedeman C, Dunn JR, Schaffner W, Paulozzi LJ, Jones TF. High-risk use by patients prescribed opioids for pain and its role in overdose deaths. JAMA Intern Med. 2014 May;174(5):796-801. doi: 10.1001/jamainternmed.2013.12711. PMID 24589873
- [Background] Gomes T, Mamdani MM, Dhalla IA, Paterson JM, Juurlink DN. Opioid dose and drug-related mortality in patients with nonmalignant pain. Arch Intern Med. 2011 Apr 11;171(7):686-91. doi: 10.1001/archinternmed.2011.117. PMID 21482846
- [Background] Paulozzi LJ, Budnitz DS, Xi Y. Increasing deaths from opioid analgesics in the United States. Pharmacoepidemiol Drug Saf. 2006 Sep;15(9):618-27. doi: 10.1002/pds.1276. PMID 16862602
- [Background] Warner M, Chen LH, Makuc DM. Increase in fatal poisonings involving opioid analgesics in the United States, 1999-2006. NCHS Data Brief. 2009 Sep;(22):1-8. PMID 19796521
- [Background] Talmi YP, Horowitz Z, Pfeffer MR, Stolik-Dollberg OC, Shoshani Y, Peleg M, Kronenberg J. Pain in the neck after neck dissection. Otolaryngol Head Neck Surg. 2000 Sep;123(3):302-6. doi: 10.1067/mhn.2000.104946. PMID 10964311
- [Background] Chen SC, Liao CT, Chang JT. Orofacial pain and predictors in oral squamous cell carcinoma patients receiving treatment. Oral Oncol. 2011 Feb;47(2):131-5. doi: 10.1016/j.oraloncology.2010.11.004. Epub 2010 Dec 13. PMID 21147547
- [Background] Bianchini C, Malago M, Crema L, Aimoni C, Matarazzo T, Bortolazzi S, Ciorba A, Pelucchi S, Pastore A. Post-operative pain management in head and neck cancer patients: predictive factors and efficacy of therapy. Acta Otorhinolaryngol Ital. 2016 Apr;36(2):91-6. doi: 10.14639/0392-100X-499. Epub 2016 Apr 29. PMID 27196072
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Background] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990
- See also: PROSPECT website — https://esraeurope.org/prospect/